CLINICAL TRIAL: NCT00890890
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Tolerability, Pharmacodynamic and Pharmacokinetic Effects of BMS-708163 in the Treatment of Patients With Prodromal Alzheimer's Disease
Brief Title: A Multicenter, Double Blind, Placebo-Controlled, Safety and Tolerability Study of BMS-708163 in Patients With Prodromal Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN156-018; 2009-010067-16 (EudraCT Number)
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — BMS 708163

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Avagacestat (50 mg) (Experimental)
  Interventions: Drug: Avagacestat
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avagacestat — Capsules, Oral, 50 mg, once daily, 104 - 220 Weeks
  Other Names: BMS-708163
  Arms: Avagacestat (50 mg)
Drug: Placebo — Capsules, Oral, 0 mg, once daily, 104 - 220 Weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and tolerability of BMS-708163 in patients with Prodromal Alzheimer's disease over a treatment period of a minimum of 104-weeks. In addition patients will be seen for safety visits at 4 and 12 weeks post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets clinical criteria for prodromal Alzheimer's disease (MMSE 24-30)
* Memory complaint by subject or study partner
* CSF aβ42 levels < 200pg/mL or Total Tau/aβ42 ratio of ≥ 0.39
* Score of ≤4 on the Modified Hachinski Ischemia Scale
* CT results consistent with Alzheimer's disease
* Medically stable
* 6 years education
* Reliable study partner
* Must be able to swallow capsules

Exclusion Criteria:

* Premenopausal women
* DSM-IV diagnosis of Dementia History of stroke
* Immunocompromised
* Active peptic ulcer, GI bleed, chronic inflammatory bowel disease, chronic diarrhea or past GI surgery that would impact drug absorption
* Unstable Vitamin B-12 deficiency
* Hematologic or solid malignancy within 5 years
* Geriatric Depression Scale ≥ 6
* Unstable medical condition
* Alcohol or drug abuse history with 12-months of study entry
* Significant drug allergy
* Prisoners, compulsory psychiatric patients, or residents of nursing home or skilled nursing facility at entry
* Any other experimental therapy with 30-days of study entry

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2009-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of BMS-708163 in patients with Prodromal Alzheimer's disease as measured by adverse events, vital signs, laboratory assessments, electrocardiograms (ECGs) and Safety Head Magnetic resonance imaging (MRI) findings | Every 12 weeks up to week 220
Safety and tolerability of BMS-708163 in patients with Prodromal Alzheimer's disease as measured by adverse events, vital signs, laboratory assessments, electrocardiograms (ECGs) and Safety Head Magnetic resonance imaging (MRI) findings | Avagacestat-treated patients will be seen for safety visits at 4 Post Treatment/Study Termination
Safety and tolerability of BMS-708163 in patients with Prodromal Alzheimer's disease as measured by adverse events, vital signs, laboratory assessments, electrocardiograms (ECGs) and Safety Head Magnetic resonance imaging (MRI) findings | Avagacestat-treated patients will be seen for safety visits at 12 Post Treatment/Study Termination
Safety and tolerability of BMS-708163 in patients with Prodromal Alzheimer's disease as measured by adverse events, vital signs, laboratory assessments, electrocardiograms (ECGs) and Safety Head Magnetic resonance imaging (MRI) findings | Avagacestat-treated patients will have a 24 week post treatment skin examination by a dermatologist

SECONDARY OUTCOMES:
Predictive value of Cerebral Spinal Fluid (CSF) biomarkers (Aβ40, and Aβ42, total Tau, total Tau/Aβ42 ratio, phosphorylated Tau) on progression to dementia | Baseline (Week 0), Week 2 (optional), Week 24 and Week 104

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (64):
- United States (50):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Pivotal Research Centers, Peoria, Arizona
  - 21st Century Neurology, Phoenix, Arizona
  - Banner Alzheimer'S Institute, Phoenix, Arizona
  - Sun Health Research Institue, Sun City, Arizona
  - Margolin Brain Institute, Fresno, California
  - Collaborative Neuroscience Network, Inc., Long Beach, California
  - Mary S. Easton Center, Los Angeles, California
  - Pharmacology Research Institute, Newport Beach, California
  - Uc Irvine Medical Center, Orange, California
  - Pacific Research Network, San Diego, California
  - Affiliated Research Institute, San Diego, California
  - University Of California, San Diego, San Diego, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - Radiant Research, Inc., Denver, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Meridien Research, Brooksville, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Md Clinical, Hallandale, Florida
  - Compass Research, Llc, Orlando, Florida
  - Indiana University Medical Center, Indianapolis, Indiana
  - Four Rivers Clinical Research, Inc, Paducah, Kentucky
  - Brigham & Women'S Hospital, Boston, Massachusetts
  - St Louis University, St Louis, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Center For Brain Health, Las Vegas, Nevada
  - Memory Enhancement Center Of Amercia, Inc., Eatontown, New Jersey
  - Robert Wood Johnson Medical School, Umdnj, New Brunswick, New Jersey
  - Global Medical Institutes, Llc, Princeton, New Jersey
  - Memory Enhancement Center Of Nj, Inc., Toms River, New Jersey
  - Spri Clinical Trials, Llc, Brooklyn, New York
  - Nyu Langone Medical Center, New York, New York
  - Columbia University, New York, New York
  - University Of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Raleigh Neurology Associates, Pa, Raleigh, North Carolina
  - Richard H. Weisler, Md, Pa & Assoc., Raleigh, North Carolina
  - Clinical Trials Of America, Inc., Winston-Salem, North Carolina
  - Wake Forest University School Of Medicine, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Neurology & Neuroscience Center Of Ohio, Toledo, Ohio
  - Tulsa Clinical Research, Llc, Tulsa, Oklahoma
  - Providence Cognitive Assessment Clinic, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Butler Hospital, Providence, Rhode Island
  - Senior Adults Specialty Research (Sasr), Austin, Texas
  - The University Of Texas, Dallas, Texas
  - Dean Foundation For Health Research & Education, Middleton, Wisconsin
  - Mcw Clinics At Froedtert Hospital, Milwaukee, Wisconsin
- Canada (5):
  - Local Institution, Calgary, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, London, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Greenfield Park, Quebec
- Local Institution, Copenhagen, Denmark
- Local Institution, Turku, Finland
- France (5):
  - Local Institution, Toulouse, Cedex 9
  - Local Institution, Bordeaux
  - Local Institution, Dijon
  - Local Institution, Nantes
  - Local Institution, Rennes
- Sweden (2):
  - Local Institution, Mölndal
  - Local Institution, Stockholm

REFERENCES:
- [Derived] Coric V, Salloway S, van Dyck CH, Dubois B, Andreasen N, Brody M, Curtis C, Soininen H, Thein S, Shiovitz T, Pilcher G, Ferris S, Colby S, Kerselaers W, Dockens R, Soares H, Kaplita S, Luo F, Pachai C, Bracoud L, Mintun M, Grill JD, Marek K, Seibyl J, Cedarbaum JM, Albright C, Feldman HH, Berman RM. Targeting Prodromal Alzheimer Disease With Avagacestat: A Randomized Clinical Trial. JAMA Neurol. 2015 Nov;72(11):1324-33. doi: 10.1001/jamaneurol.2015.0607. PMID 26414022
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx